CLINICAL TRIAL: NCT07185373
Title: Orelabrutinib Combined With Teniposide, Rituximab and Methotrexate for Newly Diagnosed Primary Central Nervous System Lymphoma-A Randomized Controlled Trial
Brief Title: Orelabrutinib Combined With Teniposide, Rituximab and Methotrexate for Newly Diagnosed PCNSL
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Tong Chen, MD, Prof., Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-725
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — Teniposide; orelabrutinib; Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Teniposide, orelabrutinib, rituximab, methotrexate (MTX), and dexamethasone (21-day cycle).
  Interventions: Drug: Teniposide; Drug: Orelabrutinib; Drug: MTX; Drug: Rituximab (R); Drug: Dexamethasone
- Arm B (Experimental): Orelabrutinib, rituximab, MTX and dexamethasone (21-day cycle).
  Interventions: Drug: Orelabrutinib; Drug: MTX; Drug: Rituximab (R); Drug: Dexamethasone
- Arm C (Active Comparator): Rituximab, MTX and dexamethasone (21-day cycle)
  Interventions: Drug: MTX; Drug: Rituximab (R); Drug: Dexamethasone

INTERVENTIONS:
Drug: Teniposide — This trial enrolls eligible participants (meeting inclusion and exclusion criteria), who will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification factors include age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.
  Induction regimens:
  Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone, administered in 21-day cycles.
  Arm B: Orelabrutinib, rituximab, MTX and dexamethasone, administered in 21-day cycles.
  Arm C: Rituximab, MTX and dexamethasone, administered in 21-day cycles. Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will proceed to consolidation therapy.
  Arms: Arm A
Drug: Orelabrutinib — This trial enrolls eligible participants (meeting inclusion and exclusion criteria), who will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification factors include age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.
  Induction regimens:
  Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone, administered in 21-day cycles.
  Arm B: Orelabrutinib, rituximab, MTX and dexamethasone, administered in 21-day cycles.
  Arm C: Rituximab, MTX and dexamethasone, administered in 21-day cycles. Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will proceed to consolidation therapy.
  Arms: Arm A; Arm B
Drug: MTX — This trial enrolls eligible participants (meeting inclusion and exclusion criteria), who will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification factors include age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.
  Induction regimens:
  Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone, administered in 21-day cycles.
  Arm B: Orelabrutinib, rituximab, MTX and dexamethasone, administered in 21-day cycles.
  Arm C: Rituximab, MTX and dexamethasone, administered in 21-day cycles. Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will proceed to consolidation therapy.
Drug: Rituximab (R) — This trial enrolls eligible participants (meeting inclusion and exclusion criteria), who will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification factors include age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.
  Induction regimens:
  Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone, administered in 21-day cycles.
  Arm B: Orelabrutinib, rituximab, MTX and dexamethasone, administered in 21-day cycles.
  Arm C: Rituximab, MTX and dexamethasone, administered in 21-day cycles. Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will proceed to consolidation therapy.
Drug: Dexamethasone — This trial enrolls eligible participants (meeting inclusion and exclusion criteria), who will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification factors include age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.
  Induction regimens:
  Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone, administered in 21-day cycles.
  Arm B: Orelabrutinib, rituximab, MTX and dexamethasone, administered in 21-day cycles.
  Arm C: Rituximab, MTX and dexamethasone, administered in 21-day cycles. Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will proceed to consolidation therapy.

SUMMARY:
This is a three-arm, multicenter, randomized controlled trial. Eligible participants will be randomized to one of three induction regimens via stratified block randomization at a 2:2:1 ratio.

Induction regimens:

Arm A: Teniposide + orelabrutinib + rituximab + methotrexate (MTX) + dexamethasone, administered in 21-day cycles.

Arm B: Orelabrutinib + rituximab + MTX + dexamethasone, administered in 21-day cycles.

Arm C: Rituximab + MTX + dexamethasone, administered in 21-day cycles. Participants achieving complete response (CR) or unconfirmed complete response (CRu) post-induction will proceed to consolidation therapy, with options including: MTX + rituximab (once every 3 months for 1 year); high-dose chemotherapy followed by autologous stem cell transplantation (ASCT); dose-reduced whole brain radiotherapy; or other modalities (as determined by the investigator).

DETAILED DESCRIPTION:
This is a three-arm, multicenter, randomized controlled trial. Eligible participants (meeting inclusion and exclusion criteria) will be assigned to one of three induction regimens via stratified block randomization at a 2:2:1 ratio. Stratification will be based on two factors: age (≤60 vs. >60 years) and ECOG performance status (0-1 vs. 2-3). Within each stratum, blocks of size 15 will be used to ensure balanced allocation.

Induction regimens:

Arm A: Teniposide, orelabrutinib, rituximab, methotrexate (MTX) and dexamethasone (21-day cycle).

Arm B: Orelabrutinib, rituximab, MTX and dexamethasone (21-day cycle). Arm C: Rituximab, MTX and dexamethasone (21-day cycle).

Following induction therapy, participants achieving complete response (CR) or unconfirmed complete response (CRu) will receive consolidation therapy. Four options are available, with selection determined by investigators based on individual patient conditions in real-world practice:

Chemotherapy (MTX + rituximab, administered once every 3 months for 1 year); High-dose chemotherapy conditioning followed by autologous stem cell transplantation (ASCT); dose-reduced whole brain radiotherapy; Other consolidation modalities. Participants who do not achieve CR or CRu after induction therapy will be eligible for alternative anti-primary central nervous system lymphoma (anti-PCNSL) treatments, as determined by investigators based on individual clinical status.

ELIGIBILITY:
Inclusion Criteria:

* No prior systemic treatment for primary central nervous system lymphoma
* Pathologically confirmed as diffuse large B-cell lymphoma subtype; with sufficient residual surgical specimens remaining after meeting the needs for pathological diagnosis and preservation
* Aged 18-75 years (inclusive)
* ECOG performance status ≤3
* Expected survival time exceeding 3 months
* Major organ functions meeting the following standards:

  1. Blood routine parameters (without growth factor support or blood transfusion within the past 7 days; 14 days for pegylated myeloid growth factors): absolute neutrophil count (ANC) ≥1.0×10⁹/L, platelet count (PLT) ≥75×10⁹/L, hemoglobin (Hb) ≥80g/L;
  2. Blood biochemistry: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) or ≤3×ULN (for confirmed Gilbert syndrome with direct bilirubin within normal range); aspartate transaminase (AST) or alanine transaminase (ALT) ≤2.5×ULN; serum creatinine within normal range; estimated glomerular filtration rate (eGFR) ≥70ml/min;
  3. Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5×ULN;
* Ability to tolerate lumbar puncture and/or having an indwelling Ommaya reservoir
* Peripheral blood flow cytometry showed no clonal B cells and no other extramedullary lesions.
* Voluntary signing of a written informed consent form by the participant or their legal representative prior to trial screening, indicating their understanding of the study purpose, necessary procedures, and willingness to comply with the protocol and attend follow-up visits

Exclusion Criteria:

* Lymphoma involving sites outside the central nervous system (CNS)
* Patients with a previous history of tumors
* Patients with intraocular lymphoma or suspected diagnosis of intraocular lymphoma invasion
* Uncontrolled or significant cardiovascular diseases, including:

  1. New York Heart Association (NYHA) class Ⅲ-Ⅳ congestive heart failure, unstable angina, myocardial infarction within 6 months prior to the first administration of study drugs; clinically significant or treatment-requiring arrhythmias at screening; left ventricular ejection fraction (LVEF) <50%; or patients with controlled coronary heart disease who are either not using anticoagulants/antiplatelet drugs or taking 2 or more anticoagulants/antiplatelet drugs orally.
  2. Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, unclassified cardiomyopathy).
  3. A history of clinically significant QTc interval prolongation, or QTc interval (calculated via Bazett's formula using manually collected screening data) >470ms in females or >450ms in males.
  4. Refractory hypertension (blood pressure not controlled despite ≥1 month of optimal, tolerable doses of 2 or more antihypertensive drugs [including diuretics] with lifestyle modifications; or blood pressure controlled only with 3 or more antihypertensive drugs).
* Active bleeding within 2 months prior to screening; use of anticoagulants/antiplatelet drugs for <6 months; or a definite bleeding tendency as judged by the investigator (e.g., bleeding-risk esophageal varices, active local ulcer lesions).
* Diabetic patients whose blood sugar remains poorly controlled after insulin treatment
* A history of stroke or intracranial hemorrhage within 6 months prior to screening, excluding postoperative sequelae-related intracranial hemorrhage
* A history of organ transplantation or allogeneic bone marrow transplantation
* Surgical procedures within 6 weeks prior to screening (diagnostic examinations are not considered surgical procedures; insertion of vascular access devices is exempt from this exclusion criterion).
* Use of Chinese herbal medicines with anti-tumor effects (as specified in the package insert, e.g., Compound Cantharidin Capsules) within 4 weeks prior to screening
* Active or uncontrolled hepatitis B virus (HBV) infection (HBsAg positive and/or HBcAb positive with positive HBV DNA titer); HCV Ab positive; HIV positive. The following patients can be provisioned for continuous observation pending enrollment when given prophylactic anti-HBV (such as entecavir or tenofovir), including :

  1. HBsAg positive with negative HBV DNA titer.
  2. HBsAg negative, HBsAb negative, HBcAb positive, and negative HBV DNA titer Patients with positive HBV-DNA can be considered for enrollment only when the HBV-DNA value is less than 500IU/mL after treatment
* Uncontrolled active systemic fungal, bacterial, viral, or other infections (defined as persistent infection-related symptoms/signs that do not improve despite appropriate antibiotic or other treatments) or requiring intravenous antibiotics
* Administration of live vaccines or immunological agents within 4 weeks prior to enrollment.
* Need for concurrent and continuous use of drugs with moderate/strong inhibitory or inductive effects on cytochrome P450 CYP3A.
* Patients with hypersensitivity to orelabrutinib or its excipients (e.g., immediate or accelerated allergic reactions).
* Patients with hypersensitivity to teniposide or its excipients (e.g., immediate or accelerated allergic reactions)
* Clinically significant gastrointestinal abnormalities that may affect drug intake, transit, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or participants with total gastrectomy.
* Participants with a history or current presence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia with severely impaired lung function, etc
* Participants with chronic liver damage, severe fatty liver, or alcoholic liver disease.
* Pregnant or lactating women; women of childbearing age who are unwilling to use contraception from the time of enrollment until 180 days after the last dose of the study drug (serum pregnancy test results must be negative within 14 days before the start of study drug treatment for women of childbearing potential); men who are not surgically sterilized and unwilling to use contraception during the study and until 180 days after the last dose of the study drug.
* Presence of life-threatening diseases or severe organ dysfunction, deemed unsuitable for participation in the trial by the investigator.
* Any mental or cognitive impairment that may limit the understanding and execution of the informed consent form or adherence to the study
* Previous receipt of whole-brain radiotherapy for primary central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of CR/CRu in Arm A versus Arm C during the induction therapy phase | At the end of Cycle6 (each cycle is 21 days)
  Efficacy evaluation will be determined in accordance with the IPCG criteria
The proportion of CR/CRu in Arm A versus Arm B during the induction therapy phase | At the end of Cycle6 (each cycle is 21 days)
  Efficacy evaluation will be determined in accordance with the IPCG criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) during induction therapy | At the end of Cycle6 (each cycle is 21 days)
  Efficacy evaluation will be determined in accordance with the IPCG criteria
proportion of CR/CRu in Arm B versus Arm C during the induction therapy phase | At the end of Cycle6 (each cycle is 21 days)
  Efficacy evaluation will be determined in accordance with the IPCG criteria
Progression-free survival (PFS) | 2 years after Day 1 Cycle 1
  Efficacy evaluation will be determined in accordance with the IPCG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Tong Chen, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - West China Hospital of Sichuan University, Chengdu
  - Department of Hematology, Qilu Hospital of Shandong University, Jinan